CLINICAL TRIAL: NCT00105586
Title: Pharmacotherapy of Late-Life Generalized Anxiety Disorder
Brief Title: Drug Therapy for Generalized Anxiety Disorder Among the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH070547 (NIH); R01MH070547 (NIH)
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder
Keywords: Anxiety; Elderly; Aged; Serotonin Reuptake Inhibitors; SSRI; SERT
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram (1) (Experimental): Escitalopram
  Interventions: Drug: Escitalopram
- Placebo (2) (Placebo Comparator): Placebo
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Participants will either take 10 to 20 mg of escitalopram or placebo. Participants who wish to participate in the open-label extension receive an additional 12 weeks of escitalopram.
  Other Names: Lexapro

SUMMARY:
This study will determine the efficacy of escitalopram (Lexapro®), an anti-anxiety drug, for generalized anxiety disorder (GAD) and the ways genetics affect response to treatment for GAD in elderly individuals.

DETAILED DESCRIPTION:
GAD is a serious public health issue; particularly among the elderly, prevalence of the condition is high, and functional burden on those with the illness is significant. GAD is associated with irregular levels of neurotransmitters, chemicals that carry messages across nerve endings. Serotonin is a neurotransmitter that helps regulate mood and emotions; increased levels of serotonin have been shown to reduce anxiety. Standard treatment for GAD typically involves selective serotonin reuptake inhibitors (SSRIs), drugs that reduce serotonin re-entry into nerve cells. Escitalopram is an SSRI that is well tolerated and highly specific for the serotonin transporter (SERT). The primary aim of this study is to examine the efficacy of escitalopram in reducing anxiety symptoms among elderly GAD patients. Additional aims include examining the efficacy of escitalopram for improving function, quality of life, and neuropsychological functioning, and examining whether genetic variation in the SERT gene influences these participants' response to treatment.

Participants will be randomly assigned to receive either escitalopram or placebo for 12 weeks (there is also a 12 week open label extension in which all participants will receive escitalopram). Participants will have weekly/biweekly study visits; during these visits, participants will complete self-report questionnaires on functional ability and anxiety symptoms. Blood collection and cognitive testing through various tasks will also occur.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least moderately severe generalized anxiety disorder (GAD)

Exclusion Criteria:

* Serious suicide risk or psychiatric instability that would affect study participation
* Dementia
* Substance abuse, such as alcoholism, within 6 months prior to study entry
* Diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or bipolar disorder
* Unstable medical conditions that would preclude the use of escitalopram
* Use of certain psychotropics that can not be safely tapered or discontinued for at least 2 weeks prior to and during the study
* Use of neuroleptics that are absorbed over a prolonged period of time within 6 weeks prior to study entry

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2004-12; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Lenze, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
interested investigators should contact the PI directly via email.

REFERENCES:
- [Result] Lenze EJ, Rollman BL, Shear MK, Dew MA, Pollock BG, Ciliberti C, Costantino M, Snyder S, Shi P, Spitznagel E, Andreescu C, Butters MA, Reynolds CF 3rd. Escitalopram for older adults with generalized anxiety disorder: a randomized controlled trial. JAMA. 2009 Jan 21;301(3):295-303. doi: 10.1001/jama.2008.977. PMID 19155456
- [Result] Butters MA, Bhalla RK, Andreescu C, Wetherell JL, Mantella R, Begley AE, Lenze EJ. Changes in neuropsychological functioning following treatment for late-life generalised anxiety disorder. Br J Psychiatry. 2011 Sep;199(3):211-8. doi: 10.1192/bjp.bp.110.090217. Epub 2011 Jul 4. PMID 21727232
- [Derived] Altmann H, Stahl ST, Gebara MA, Lenze EJ, Mulsant BH, Blumberger DM, Reynolds CF 3rd, Karp JF. Coprescribed Benzodiazepines in Older Adults Receiving Antidepressants for Anxiety and Depressive Disorders: Association With Treatment Outcomes. J Clin Psychiatry. 2020 Sep 29;81(6):20m13283. doi: 10.4088/JCP.20m13283. PMID 32991792
- [Derived] Lenze EJ, Goate AM, Nowotny P, Dixon D, Shi P, Bies RR, Lotrich FK, Rollman BL, Shear MK, Thompson PA, Andreescu C, Pollock BG. Relation of serotonin transporter genetic variation to efficacy of escitalopram for generalized anxiety disorder in older adults. J Clin Psychopharmacol. 2010 Dec;30(6):672-7. doi: 10.1097/jcp.0b013e3181fc2bef. PMID 21105279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 257 subjects consented (177 randomized and received treatment)
Pre-assignment Details: 78 excluded from randomization due to ineligibility and/or refusal; 2 excluded after randomization but did not start treatment
Groups:
- Placebo: Participants will receive a placebo.
- Escitalopram: Participants will receive escitalopram.
Period: Overall Study
Arm/Group | Placebo | Escitalopram
Started | 92 | 85
Completed | 75 | 69
Not Completed | 17 | 16
Not completed — Adverse Event | 4 | 3
Not completed — Physician Decision | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Escitalopram | Total
Number analyzed (Participants) | 92 | 85 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 92 | 85 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (8.2) | 71.1 (7.4) | 71.6 (9.9999)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 34 | 24 | 58
Region of Enrollment [Number; unit: participants]
  United States | 92 | 85 | 177.0

OUTCOME MEASURES:

1. Primary Outcome: Response Using Clinical Global Impressions-Improvement Scale (CGI-I)
Description: Cumulative incident response of anxiety symptom improvement on CGI-I, with 1 (very much improved) to 2 (much improved) indicated as response. Scores synthesized from anxiety rating scale scores, including Penn State Worry Questionnaire (PSWQ) and Hamilton Anxiety Scale (HamA).
Time Frame: Measured at Weeks 1-12
Measure: Number; unit: participants
Arm/Group | Placebo | Escitalopram
Number analyzed (Participants) | 75 | 69
participants | 51 | 69

2. Secondary Outcome: Quality of Life
Description: Role -emotional impairment score from the Late-Life Function and Disability Instrument (min score=0, significant impairment; max score=100, no impairment).
Time Frame: Measured at Week 12
Population: Quality of Life scales were collected on all participants randomized to Escitalopram and placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram (1) | Placebo (2)
Number analyzed (Participants) | 85 | 92
units on a scale
  Week 0 SF-36 Role-Emotional Impairment | 42.19 (36.72) | 53.42 (38.39)
  Week 12 SF-36 Role-Emotional Impairment | 62.50 (37.80) | 56.16 (38.83)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/85
Other Adverse Events (participants affected / at risk) | 59/92 | 65/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | Escitalopram (N=85)
Fatigue or somnolence (General disorders) | 10 | 25
Gastrointestinal upset (Gastrointestinal disorders) | 26 | 22
Headache (General disorders) | 7 | 13
Sleep disturbance (General disorders) | 2 | 12
Sweating (Nervous system disorders) | 5 | 11
Urinary symptoms (Renal and urinary disorders) | 0 | 8 — increased or decreased frequency and urgency
Increased anxiety or depression (Psychiatric disorders) | 9 | 7
Light-headedness (Nervous system disorders) | 7 | 7
Tremor (Nervous system disorders) | 2 | 7
Aches (Musculoskeletal and connective tissue disorders) | 14 | 5
Rash or pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Sexual (Reproductive system and breast disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less